CLINICAL TRIAL: NCT06512233
Title: Dual Therapy Dilemma: Heparin Alone vs. Heparin-Aspirin Combo in Free Flap Survival
Brief Title: Heparin Alone vs. Heparin-Aspirin Combo in Free Flap Survival
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Aga Khan University (Other)
Responsible Party: Principal Investigator, Ceemal Khan, Research Associate, Aga Khan University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 000000
Record Dates: First submitted 2024-07-16; First posted 2024-07-22 (Actual); Last update posted 2024-07-23 (Actual); Status verified 2024-07

CONDITIONS: Complication,Postoperative
Keywords: Ischemia; Thrombosis; Vascular Complications; Surgical Wound Healing; Reconstructive Surgery Complications
MeSH Terms: conditions — Postoperative Complications; Ischemia; Thrombosis | interventions — Dalteparin; Aspirin

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- LMW Heparin 5000 U/ML-Aspirin 75 MG (Active Comparator): Patients will receive 5000 unit of low molecular weight heparin subcutaneously once daily along with tablet aspirin 75 MG once daily, for additional thromboprophylaxis for free flap. The flaps of these patients will be monitored as standard clinical examination and outcome will be recorded until 4th post operative day.
  Interventions: Drug: LMW Heparin 5000 U/ML-Aspirin 75 MG
- LMW Heparin 5000 U/ML (Active Comparator): Patients will receive 5000 unit of low molecular weight heparin subcutaneously once daily according to institutional protocol as routine practice for prevention of deep venous thrombosis in post operative period. The flaps of these patients will be monitored as standard clinical examination and outcome will be recorded until 4th post operative day.
  Interventions: Drug: LMW Heparin 5000 U/ML

INTERVENTIONS:
Drug: LMW Heparin 5000 U/ML-Aspirin 75 MG — Arm 1
  Arms: LMW Heparin 5000 U/ML-Aspirin 75 MG
Drug: LMW Heparin 5000 U/ML — Arm 2
  Arms: LMW Heparin 5000 U/ML

SUMMARY:
This randomized clinical trial aims to compare the effectiveness of heparin alone versus combination therapy of Heparin- Aspirin in improving free flap survival in patients undergoing reconstructive surgery. Participants will be randomly assigned to receive either heparin or a combination therapy, and the primary outcome measure will be the survival rate of the free flap at various time points post-surgery

DETAILED DESCRIPTION:
The objective of this randomized clinical trial is to evaluate the efficacy of heparin alone vs compared to combination therapy of Heparin-Aspirin in enhancing free flap survival in patients undergoing reconstructive surgery. Participants will be randomly assigned to one of two groups: one receiving standard heparin therapy and the other receiving a combination therapy that includes heparin and other agents. The primary outcome will be the survival rate of the free flap, assessed at multiple intervals after surgery. Secondary outcomes will to assess the incidence of flap thrombosis, bleeding complications, re-operation in free flap surgeries and overall patient outcomes in both groups. Ethical approval will be obtained, and informed consent will be required from all participants. This trial seeks to provide robust evidence on the potential benefits of combination therapy over heparin alone in free flap survival, potentially informing future clinical guidelines.

ELIGIBILITY:
Inclusion Criteria:

* Patients undergoing free flap surgery
* Age between 18 and 70 years

Exclusion Criteria:

* Known hypersensitivity to heparin or aspirin
* History of bleeding disorders
* Concurrent use of other anticoagulant or antiplatelet medications
* Severe renal or hepatic impairment
* Preoperative use of aspirin that could not be stopped five days before surgery due to a higher risk of cardiac-related complications.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 126 (Estimated)
Dates: Start 2025-01 (Estimated); Primary Completion 2025-12 (Estimated); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
Free Flap Survival Rate | two hourly for 1st 24 hours and then three hourly for next 48 hours and four hourly for next 72 hours and onwards.
  Percentage of patients with successful survival of the free flap grafts at specified time points post-surgery

SECONDARY OUTCOMES:
flap thrombosis, bleeding complications, re-operation in free flap surgeries and overall patient outcomes in both groups | 30 days post-surgery
  Number of participants experiencing complications requiring medical or surgical intervention within the first 30 days post-surgery.

CONTACTS AND LOCATIONS:
Overall Officials: Fizzah Arif, MD, Principal Investigator — Aga Khan University; Fazlur Rahman, MD, Study Director — Aga Khan University
Locations (1):
- Aga Khan University, Karachi, Sindh, Pakistan

IPD SHARING:
Plan to Share IPD: No